CLINICAL TRIAL: NCT03371446
Title: Effect of Smoking on the DNA Methylation Profile of the SOCS 1 Gene Promoter in Oral Mucosal Epithelial Cells of Individuals With Chronic Periodontitis (Smokers and Nonsmokers).
Brief Title: DNA Methylation Profile of the SOCS-1 Gene Promoter in Smokers Patients With Chronic Periodontitis.
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Teacher of Periodontia- Department of Buco Maxillofacial Surgery and Traumatology and Periodontics, University of Sao Paulo
Other Study IDs: CAAE: 57171816.2.0000.5419
Record Dates: First submitted 2017-11-30; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Periodontal Diseases; Epigenetics
Keywords: DNA Methylation. Smoking. SOCS-1 gene.
MeSH Terms: conditions — Periodontal Diseases | interventions — Sucrose

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — ephitelials cells of oral mocose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smokers/Non-smokers: It was an experimental study with parallel controls, comparing two groups, a group with patients who smoked for more than 10 years, consuming 10 more cigarettes per day and diagnosing chronic periodontitis (case) and another group (control) were non-smokers with chronic periodontitis, according to the standard of World Health Organization (WHO) definition of the smoking population
  Interventions: Genetic: oral epithelial cells obtained by rinsing with 3% sucrose

INTERVENTIONS:
Genetic: oral epithelial cells obtained by rinsing with 3% sucrose — rinsing with 3% sucrose, for a single time of collection, patients received periodontal treatment after collection and data analysis.

SUMMARY:
Periodontitis is related to host genetics, constitution of the dental biofilm and environmental factors such as smoking. DNA methylation is a mechanism of genetic expression that can inhibit or silence gene expression. In this way several researchers have been dedicated to study the genetic influence on the susceptibility and / or increased risk to periodontal disease. Studies have reported association between several epigenetic biomarkers with periodontal inflammation. Considering the hypothesis that there is an association between smoking and methylation in genes related to periodontal disease, the objective of this study was to verify the DNA methylation pattern in oral epithelial cells of patients with chronic periodontitis (CP) in the promoter of a specific gene involved in the control of inflammation, as suppressor of cytokine signaling (SOCS) 1 in smokers and nonsmokers patients.

DETAILED DESCRIPTION:
This was an experimental type study with parallel controls, comparing two groups, a group with consumption of 10 minimum cigarettes per day, with a diagnosis of chronic periodontitis. And another control group were non-smokers with chronic periodontitis. For this, genomic DNA was purified from oral epithelial cells obtained by rinsing with 3% sucrose, for a single time of collection, patients received periodontal treatment after collection and data analysis. The DNA was modified by Sodium bisulfite and the methylation patterns of the DNA were analyzed with the MSPCR technique (Polymerase chain reaction). This study was approved by the Institutional Review Board of the School of Dentistry of Ribeirão Preto (CAAE:57171816.2.0000.5419 ), and all patients need to provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Periodontitis carriers - presence of proximal insertion loss ≥5 mm in more than 30% of the teeth present.
* Periodontal pocket ≥ 5mm
* Smokers who have smoked 10 or more cigarettes per day for the past five years.
* No positive history of basic periodontal treatment in the last six months.

Exclusion Criteria:

* Extensive prosthetic involvement.
* Using anti-inflammatories.
* Pregnant or nursing.
* Presence of systemic alterations that compromise host response or require prophylactic medication for treatment.
* History of constant use of oral antiseptics in the last six months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who smoked for more than 10 years, consuming 10 more cigarettes per day and diagnosing chronic periodontitis (case) and another group (control) were non-smokers with chronic periodontitis, according to the standard of WHO definition of the smoking population,The ChP was diagnose in accordance with the recommended standards from the Center for Disease control and Prevention, the American Academy of Periodontology on the condition of patients in good general health, aged over 30 years, presenting with pocket periodontal disease with CAL ≥ 5 mm and radiographic bone loss and bleeding after probing.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-11-18 (Actual)

PRIMARY OUTCOMES:
Extraction of genomic DNA from oral epithelial cells | Baseline (at the beginning of the study)
  Epithelial cells were collected after mouthwash with 5ml dextrose autoclaved 3% and stored under refrigeration at -20ºC. After collection, the samples were taken to the Epigenetics and Reproduction Laboratory of the Department of Genetics of the Medical School of Ribeirão Preto-USP (FMRP-USP) where nucleic acid extraction and molecular analysis were performed.
  After thawing the saliva, 2ml of each sample collected were transferred separately to eppendorf tubes, for processing. The material was then diluted in 50 μl of cobalt Mili-Q water, incubated at 37 ° C in a water bath for 1 hour and stored in a freezer at -20 ° C. At the end, DNA quality, purity and integrity were measured using a spectrophotometer (NanoDrop 2000-Thermo Scientific), using OD 260/280 and 260/230. Considering ideal values for both reasons, between 1.8 and 2.2.

SECONDARY OUTCOMES:
Probing pocket depth (PD) | Baseline (at the beginning of the study)
  Clinical parameter was recorded at baseline by one trained periodontist.Probing pocket depth (PD) was measured from the free gingival margin to the bottom of the periodontal pocket and clinical attachment level ( CAL) was measured from the cementum-enamel junction (CEJ) to the bottom of periodontal pocket.
  Probing measurement was performed using a manual University of North Carolina - UNC Periodontal probe (Hu- Friedy, Chicago, IL, USA).
Plaque index (PI) | Baseline (at the beginning of the study)
  Clinical parameter was recorded at baseline by one trained periodontist. Plaque index (PI) was used to assess the oral hygiene status of the patients, the evaluation was done with the unit of measure in percentage (%) whole mouth. Probing measurement was performed using a manual University of North Carolina - UNC Periodontal probe (Hu- Friedy, Chicago, IL, USA).
Bleeding on probing (BOP) | Baseline (at the beginning of the study)
  Clinical parameter was recorded at baseline by one trained periodontist.Bleeding on probing (BOP) was recorded based on the presence or absence of bleeding up to 30 seconds after probing on four sides of each tooth,the evaluation was done with the unit of measure in percentage (%) whole mouth. Probing measurement was performed using a manual University of North Carolina - UNC Periodontal probe (Hu- Friedy, Chicago, IL, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur B. Novaes Junior, DDS, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Arthur Belem Novaes Junior, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available with conclusion of study.
Supporting Information: Study Protocol
Time Frame: Data will be available within 2 years of study completion
Access Criteria: Data access criteria will be reviewed by the an external independent review panel.